CLINICAL TRIAL: NCT06149130
Title: Adebrelimab Combined With Dalpiciclib and Standard Endocrine Therapy for HR+/HER2 - Advanced Breast Cancer:a Single-arm, Phase II Exploratory Clinical Study
Brief Title: Adebrelimab Combined With Dalpiciclib and Standard Endocrine Therapy for HR+/HER2 - Advanced Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Huihua Xiong, Tongji Hospital Affiliated of Tongji Medical College Huazhong University of Science and Technology, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB20231105
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: HR+/HER2- breast cancer; adebrelimab; dalpiciclib
MeSH Terms: conditions — Breast Neoplasms | interventions — dalpiciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): 1. Adebrelimab: 1200mg intravenously ,Q3W
  2. dalpiciclib : 150mg once a day for 3 weeks, stop for 1 week, Q4W
  3. Endocrine recommended drugs untreated: aromatase inhibitors (letrozole/anastrozole/exemestane), given orally once daily at a specific dose (letrozole 2.5mg/ day; Anastrozole 1mg/ day, exemestane 25mg/ day); first-line endocrine therapy failed: fluvestrant was given once every 28 days, 500mg intramuscular injection, and then 500mg intramuscular injection 2 weeks after the first administration;
  Interventions: Drug: Adebrelimab; Drug: dalpiciclib

INTERVENTIONS:
Drug: Adebrelimab — adebrelimab:1200mg intravenously, Q3W.
  Other Names: SHR-1316
Drug: dalpiciclib — dalpiciclib:150mg once a day for 3 weeks and stop for 1 week. Q4W.
  Other Names: SHR-6390

SUMMARY:
This is a prospective, single-arm, multicenter Phase II study of patients with advanced HR+/HER2- breast cancer who are untreated or have failed previous first-line endocrine therapy。The primary objective of this study was to explore the efficacy and safety of the PD-L1 inhibitor adebrelimab in combination with the CDK4/6 inhibitor Dalpiciclib and standard endocrine therapy in advanced HR+/ HER2-breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal/perimenopausal or postmenopausal women aged ≥18 years and ≤75 years;
2. Histologically confirmed HR+/HER2- invasive breast cancer (specific definition: ER >10% tumor cell positive is defined as ER positive, PR >10% tumor cell positive is defined as PR positive, ER and/or PR positive is defined as HR positive; HER2 0-1+ or HER2 ++ but negative by FISH test, no amplification, defined as HER2 negative);
3. Locally advanced breast cancer (radical local treatment is not possible) or recurrent metastatic breast cancer;
4. Did not receive any systemic anti-cancer therapy at the stage of recurrence and metastasis or failed to receive first-line endocrine therapy at the advanced stage;
5. Allowed to receive ≤1 line of chemotherapy
6. Have at least one measurable lesion according to RECIST version 1.1
7. Adequate hematology and organ function, including:

   hemoglobin > 9 g/dL without blood transfusion or erythropoietin in the past 14 days.

   ANC ≥ 1.5×109/L without using granulocyte colony stimulating factor in the past 14 days.

   PLT ≥ 75×109/L without blood transfusion in the past 14 days. TBIL ≤ 1.5 ×ULN (Gilbert syndrome allows ≤ 3 × ULN). ALT and AST ≤ 3 × ULN (if there is liver metastasis, ALT and AST ≤ 5 × ULN). Serum Cr ≤ 1.5 × ULN or endogenous creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula)
8. ECOG score 0 or 1, and life expectancy ≥3 months;
9. Fertile female subjects are required to use a medically approved contraceptive during the study treatment period and for at least 3 months after the last use of the study drug;
10. Subjects voluntarily joined the study, signed informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Previous use of CDK4/6 inhibitors or PD1/PD-L1 monoclonal antibody
2. Uncontrolled central nervous system metastasis (meaning symptoms or the use of glucocorticoids or mannitol to control symptoms);
3. A history of clinically significant or uncontrolled heart disease, including congestive heart failure, angina pectoris, myocardial infarction within the last 6 months, or ventricular arrhythmia;
4. Radiotherapy, surgery, or other targeted and immunotherapy for advanced HR+/HER2- breast cancer within 4 weeks prior to first administration of the study drug;
5. Pregnant or lactating patients;
6. Malignant tumors within the past three years (except for cured basal cell carcinoma of the skin and cervical carcinoma in situ);
7. Significant comorbidities, including mental illnesses that the investigator believes will adversely affect the patient's participation in the study;
8. Those who have received anti-tumor vaccine or have received live vaccine within 4 weeks before the first administration of the investigational drug;
9. Patients with known HBV or HCV infection active phase or HBV DNA≥500, or chronic phase with abnormal liver function;
10. History of active autoimmune disease (such as interstitial pneumonia, colitis, hepatitis, pituitaritis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes)
11. A history of immunodeficiency, including HIV testing positive, or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation and allogeneic bone marrow transplantation; History of interstitial lung disease (except radiation pneumonia without hormone therapy) and non-infectious pneumonia;
12. Patients with active infection or who had been treated with systemic immune stimulating factors within 4 weeks prior to enrollment;
13. Allergic physique, or known allergic history of the drug components of this program; Or allergic to other monoclonal antibodies;
14. Previous thyroid dysfunction;
15. The investigator did not consider the patient suitable for participation in any other conditions of the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | Up to 3 years
  PFS is defined as the time from enrollment to the first imaging disease progression or death (whichever occurs first). Assessed according to RECIST v1.1 by investigator.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  ORR is defined as the proportion of patients with complete response(CR) and partial response(PR) assessed by the investigator in accordance with the RECIST 1.1 criteria.
Overall survival (OS) | Up to 5 years
  OS is defined as the time between enrollment and the patient's death due to any OS is defined as the time between enrollment and the patient's death due to any cause
Incidence of Treatment-Emergent Adverse Events | Up to 3 years
  Includes the Treatment-Emergent adverse event profile and rates according to the Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided